CLINICAL TRIAL: NCT02679352
Title: A Multicentre, Prospective Clinical Study Analysing Outcomes of Shoulder Arthroplasty with SMR STEMLESS
Brief Title: SMR Stemless Shoulder Arthroplasty Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-08
Record Dates: First submitted 2016-01-29; First posted 2016-02-10 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Primary Osteoarthritis; Secondary Osteoarthritis; Post-traumatic; Arthrosis; Rheumatoid Arthritis; Avascular Necrosis of the Head of Humerus; Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SMR stemless (Experimental): Patients requiring a primary anatomic or reverse shoulder arthroplasty, due to symptomatic painful degenerative joint diseases with good bone stock
  Interventions: Device: SMR Stemless

INTERVENTIONS:
Device: SMR Stemless — Total anatomic or reverse shoulder arthroplasty

SUMMARY:
Shoulder arthroplasty is a reliable procedure for the treatment of severe shoulder joint diseases to relieve pain and restore shoulder function.

Shoulder implants commonly used are characterised by a humeral stem and complications related to the stem are not infrequent. These include: bone stock loss, intraoperative and postoperative break around the implant, malpositioning of the humeral component and difficult eradication of infections inside the bone around the implant.

With the aim of reducing stem-related complications, a novel prosthesis characterised by a stem-less design has been developed.

The objective of this study is therefore to explore how well people recover after shoulder replacement with this novel stem-less shoulder prosthesis. This will be assessed over 5 years in three different countries in Europe using patient completed questionnaires and clinical and radiographic assessments.

DETAILED DESCRIPTION:
The hypothesis at the base of the study is that the SMR stemless system might contribute to ensure good clinical outcomes and an effective stability and might avoid the potential complications associated with a traditional stemmed implant.

The aim of this study is to assess clinical, radiographic and subjective outcomes after anatomic or reverse shoulder arthroplasty with a SMR stemless prosthesis, define the survivorship of the implant and identify possible risk factors that may lead to failure.

This is a post-marketing clinical study, because the study device is registered, CE marked and used according to the intended use.

It is an international, multi-centre, prospective case series. The assignment of any patient involved in the study is determined by the aetiology preoperatively evaluated by the Investigator and falls within current practice. The decision to use a specific prosthesis design is decided by the Investigators independently and clearly separated from the decision to include the patient in the study.

The evaluation has an internal control because the assessment of post-surgery data is compared to baseline measurements (pre-operative clinical analysis and radiographic analysis at discharge). It is open label.

The investigation will be carried out in 3 sites in Europe for a maximum total number of 78 treated patients. Accrual will be competitive until the required recruitment target is met. Equal numbers will be recruited at each of three centres (26 patients per site), but a deviation of 8 participants will be accepted (minimum of 18 and maximum of 34 participants recruited per site).

ELIGIBILITY:
Patients meeting all the following inclusion criteria will be considered for participation in the study:

1. Both genders;
2. Age ≥ 18 years old;
3. Full skeletal maturity;
4. Life expectancy over 5 years;
5. Patient is requiring primary unilateral or bilateral anatomic or reverse arthroplasty based on physical examination and medical history;
6. Good bone quality evaluated by the Investigator on the basis of a risk factors analysis (included MORES/SCORE questionnaires) and the intraoperative evaluation;
7. A diagnosis in the target shoulder of one or more of the following:

   * Primary osteoarthritis;
   * Secondary osteoarthritis;
   * Post-traumatic arthritis;
   * Rheumatoid arthritis;
   * Avascular necrosis of the humeral head (radiologically less than 20%);
   * Cuff tear arthropathy.
8. Patient submitted to previous conservative non-surgical treatments;
9. Patient is willing and able to complete scheduled follow-up evaluations as described in the Patient Information Sheet;
10. Patient has participated in the Informed Consent process and has signed the Informed Consent form previously approved by the Ethics Committee.

Patients will be excluded if they meet any of the following criteria:

1. Patient requiring revision shoulder arthroplasty;
2. Osteoporosis with a history of non-traumatic fractures;
3. Steroid injections within the previous 3 months;
4. Contralateral shoulder replacement within the previous 3 months;
5. Extensive avascular necrosis (radiologically more than 20%);
6. Meta-epiphyseal bony defect (including large cysts);
7. Post-traumatic tuberosity non-union;
8. Ongoing septicaemia;
9. Significant proven or suspicious infection of the target shoulder or any serious infectious disease before the study according to the Investigator;
10. Significant neurological or musculoskeletal disorders that may compromise functional recovery;
11. Not recovered axillary nerve palsy;
12. Non functioning deltoid muscle;
13. Known or suspicious hypersensitivity to the metal or other components and materials of the implant;
14. Recurrent medical history of immune-mediated reactions or other systemic immune disorders;
15. Current treatment or treatment for any malignancy within the previous 2 years before the preoperative visit;
16. Previous organ transplant;
17. Any intercurrent chronic disease or condition and any significant finding that may interfere with the completion of the 60-month follow-up, such as liver disease, severe coronary disease, or other clinically significant condition that the Investigator feels may affect the study evaluation;
18. Unwillingness or inability (alcoholism, infirmity) to comply with rehabilitation and to return for follow-up visits and any psychiatric illness that would prevent comprehension of the details and nature of the study;
19. Participation in any experimental drug/device study within the 6 months prior to the preoperative visit;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Efficacy as assessed by proportion of patients reaching a clinical progression measured as Constant score change | 24 months
  Constant score change of greater than 10 points

CONTACTS AND LOCATIONS:
Locations (4):
- St. Anna Hospital, Herne, Germany
- Netherlands (2):
  - Spaarne Hospital, Hoofddorp
  - Zorgsaam Zorggroep Ziekhenhuis Terneuzen, Terneuzen
- North Bristol NHS, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No